CLINICAL TRIAL: NCT00341939
Title: Retrospective Analysis of Drug Disposition and Response-related Genotypes in Cancer Patients and Correlation With Pharmacokinetics and Pharmacodynamics Data
Brief Title: Retrospective Analysis of a Drug-Metabolizing Genotype in Cancer Patients and Correlation With Pharmacokinetic and Pharmacodynamics Data
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904279; 04-C-N279
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer; Breast Cancer; Cutaneous T-Cell Lymphoma; Lung Cancer; Melanoma
Keywords: Drug Therapy; Pharmacogenetics; Cancer; Pharmacodynamics; Pharmacokinetics; Natural History
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Lymphoma, T-Cell, Cutaneous; Lung Neoplasms; Melanoma; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Cancer Patients: Cancer patients previously enrolled on IRB approved clinical trials at NCI

SUMMARY:
This study is a retrospective one, exploring the hypothesis that a person's genotypic makeup may be associated with a clinical response or toxic effect to a drug. Genetic polymorphisms, that is, states of being able to assume different forms, that are in drug-metabolizing enzymes, transporters, and receptors may affect a patient's response to drug therapy. To date, there have been limited studies looking at a drug-metabolizing genotype (genetic makeup) or phenotype (result of the genotype's interaction with the environment). However, it is often wondered if the variations in a drug's action, that is, pharmacokinetic effect, come from the genotype phenotype relationship.

Participants who entered previous clinical trials at the National Cancer Institute, as approved by the Central Institutional Review Board, may be eligible for this study. Studies for which pharmacokinetic analyses were or are being performed will be the source of the patient population.

Genotyping experiments will be performed through genomic DNA isolated from stored frozen serum. The genotyping results will be compared with pharmacokinetic data and clinical outcomes. Clinical data will consist of what is obtained during the course of the principal pharmacokinetic study. The results of the retrospective analyses will provide no direct benefit to the participants.

DETAILED DESCRIPTION:
Background

Genetic polymorphisms in drug-metabolizing enzymes, transporters/receptors, and transcription factors might affect an individual s response to drug therapy.

Inter-individual differences in efficacy and toxicity of cancer chemotherapy are especially important given the narrow therapeutic index of these drugs.

During analysis of investigational agents, inter-individual variances in pharmacokinetics and pharmacodynamics are often noted. It is often wondered if these variances might in part be explained by genetic differences in drug metabolizing enzymes, transporters, or other critical regulators of gene expression.

Objectives

To better understand the genotype-phenotype relationship, additional analysis correlating pharmacokinetic data with relevant genotyping.

Eligibility

All individuals previously enrolled on IRB approved clinical trials at the National Cancer Institute.

Design

In these retrospective studies, the association between an individual s pharmacokinetic profile and the genetic variation in their drug metabolizing enzymes and other critical regulators of gene expression will be investigated.

The hypothesis that an individual s genotypic constitution may be associated with clinical response and/or toxicity will be explored.

ELIGIBILITY:
* INCLUSION CRITERIA:

In this retrospective study, any cancer patients entered on IRB approved clinical trials at the National Cancer Institute are eligible. Studies for which pharmacokinetic analyses were/are being performed will be the source of the patient population. At this time enrollment will be limited to patients with pharmacokinetic samples obtained during treatment on protocol 00-C-0033, 00-C-0080, 01-C-0049, 01-C-0124, 01-C-0215, 02-C-0061, 02-C-0083, 02-C-0130, 02-C-0149, 02-C-0215, 02-C-0218, 02-C-0229, 03-C-0030, 03-C-0157, 03-C-0176, 03-C-0284, 04-C-0132, 04-C-0257, 04-C-0262, 04-C-0273, 04-C-0280, 05-C-0022, 05-C-0049, 05-C-0167, 05-C-0186, 06-C-0083, 06-C-0088, 06-C-0164, 06-C-0221, 07-C-0047, 07-C-0059, 07-C-0106, 07-C-0107, 08-C-0030, 08-C-0074, 94-C-0169, 95-C-0015, 97-C-0135, 97-C-0171, and 98-C-0015.

EXCLUSION CRITERIA:

A patient will be excluded if there is an insufficient quantity of sample available to perform the genotyping procedure. This is not anticipated to be of significance for this study since the methodology does not require a large serum sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals previously enrolled on IRB approved clinical trials at NCI.
Sampling Method: Non-Probability Sample
Enrollment: 484 (Actual)
Dates: Start 2004-09-07; Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the association between pharmacokinetic data and polymorphisms in drug-metabolizing enzymes and transporters | duration of study
  To retrospectively evaluate the association between pharmacokinetic data and polymorphisms in drug-metabolizing enzymes and transporters

SECONDARY OUTCOMES:
Evaluate the variability in toxicity and/or response to anticancer agents | duration of study
  To retrospectively evaluate the variability in toxicity and/or response to anticancer agents (phenotype)
Evaluate the association between new and previously identified polymorphisms (genotypes) in drug metabolism, drug targets and genes that might affect drug response | duration of study
  To retrospectively evaluate the association between new and previously identified polymorphisms (genotypes) in drug metabolism, drug targets and genes that might affect drug response

CONTACTS AND LOCATIONS:
Overall Officials: William D Figg, Pharm.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States